CLINICAL TRIAL: NCT01130935
Title: A National, Multicentre, Open-label, Non-comparative, Non-interventional Survey Examining the Frequency and Severity of Acid Related Symptoms While Taking Nexium
Brief Title: Survey Examining the Frequency and Severity of Acid Related Symptoms While Taking Nexium
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca Albania
Other Study IDs: NIS-GAL-NEX-2010/1
Record Dates: First submitted 2010-05-20; First posted 2010-05-26 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Gastric Acid Suppression; Proton Pump Inhibitors
Keywords: GERD; gastric and duodenal ulcers; NSAID therapy
MeSH Terms: conditions — Gastroesophageal Reflux; Duodenal Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This study will assess the effectiveness of Nexium at alleviating upper GI symptoms in subjects and evaluate with which treatment regimen and on which indications acid suppression with isomeric proton pump inhibitor is used in routine clinical practice in Albania.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have had upper GI symptoms requiring acid suppression treatment
* Treatment with Nexium is in accordance with indications and dosing approved in Albania.
* Start of treatment at least 2 weeks prior to enrollment to this study 5. Written informed consent is signed.

Exclusion Criteria:

* Known hypersensitivity to Nexium or any other constituents of the formulation
* Concomitant administration of atazanavir and nelfinavir.
* Alarming upper GI symptoms (i.e. significant unintended weight loss, vomiting, dysphasia, hematemesis, melena, fever, jaundice or any other sign indicating serious or malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female subjects, age > 18 years, having had upper GI symptoms requiring acid suppression treatment.
Sampling Method: Probability Sample
Enrollment: 491 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of upper GI symptoms and the overall patient's discomfort during the last week. | Day 0
Frequency and severity of upper GI symptoms and the overall patient's discomfort during the last week. | Week 2-4
Frequency and severity of upper GI symptoms and the overall patient's discomfort during the last week. | Weeks 8-12

SECONDARY OUTCOMES:
To follow the frequency, type and severity of symptoms in subjects consulting the doctors with upper GI symptoms. | Day 0
Evaluate with which treatment regimen and on which indications acid suppression with isomeric proton pump inhibitor is used in routine clinical practice in Albania. | Once: Day 0
Evaluate the tolerability of Nexium in patients with upper GI symptoms by the number of participants with adverse events. | Day 0
To follow the frequency, type and severity of symptoms in subjects consulting the doctors with upper GI symptoms. | Weeks 2-4
To follow the frequency, type and severity of symptoms in subjects consulting the doctors with upper GI symptoms. | Weeks 8-12
Evaluate the tolerability of Nexium in patients with upper GI symptoms by the number of participants with adverse events. | Weeks 2-4
Evaluate the tolerability of Nexium in patients with upper GI symptoms by the number of participants with adverse events. | Weeks 8-12

CONTACTS AND LOCATIONS:
Overall Officials: Karin Otter, MD, PhD, Study Director — Medical Director BBC; Senka Riza, Study Chair — Medical and Regulatory Manager; Skerdi Prifti, Asc.Proff., Principal Investigator — University Hospital Center "Mother Teresa"
Locations (14):
- Albania (14):
  - Research Site, Berat
  - Research Site, Burrel
  - Research Site, Durrës
  - Research Site, Elbasan
  - Research Site, Fier
  - Research Site, Kavajë
  - Research Site, Korçë
  - Research Site, Krujë
  - Research Site, Lezhë
  - Research Site, Lushnjë
  - Research Site, Peshkopi
  - Research Site, Shkodër
  - Research Site, Tirana
  - Research Site, Vlorë